CLINICAL TRIAL: NCT02049918
Title: De-identified Residual Sample Collection for the Respiratory Viral Panel on the GenMark Sample to Answer Platform (ARM 1)
Brief Title: Residual Sample Collection for Respiratory Viral Panel
Status: Completed | Type: Observational
Sponsor: GenMark Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: CTP0006
Record Dates: First submitted 2014-01-23; First posted 2014-01-30 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Respiratory Viral Illnesses: Influenza A/B, RSV, Adenovirus
Keywords: Respiratory viruses
MeSH Terms: conditions — Adenoviridae Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Nasopharyngeal Swab
Oversight: Data Monitoring Committee: No

SUMMARY:
Collect de-identified, residual samples to support a clinical trial. Samples may be prospectively or retrospectively collected. Overall Study Objective Obtain clinical performance data to characterize clinical performance of the Respiratory Viral Panel on the GenMark Sample-to-Answer Platform.

DETAILED DESCRIPTION:
The purpose of this investigational study is to collect clinical samples to establish the clinical performance characteristics of the in vitro diagnostic (IVD) Respiratory Viral Panel on the GenMark Sample-to-Answer Platform. Data obtained from the samples will be used to support premarket submissions/registrations for this GenMark product. Samples will be aliquotted, characterized by comparator methods and banked until the instrument and assay are available for testing.

Sample collection may be prospective or retrospective. Prospective collection will preserve prevalence. Retrospective collection will be used to obtain sufficient numbers of certain sample types such as where the organism of interest is of low prevalence. The Sponsor will ensure that information identifying samples as prospectively or retrospectively collected is documented.

ELIGIBILITY:
Inclusion Criteria:

* Sample from patients exhibiting signs/symptoms of respiratory viral infection
* All medical standard-of-care testing requested by the submitting clinician is complete and has been reported to the clinician/requestor.

Exclusion Criteria:

* Samples that are incorrectly de-identified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults of any age suspected of having respiratory infection.
Sampling Method: Probability Sample
Enrollment: 1487 (Actual)
Dates: Start 2013-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Sample collection study only | prospective and retrospective sample collection
  This is an IVD Diagnostic study.

CONTACTS AND LOCATIONS:
Overall Officials: Wallace Green, PhD, Principal Investigator — Milton S. Hershey Medical Center; Michelle Fennell, MHA, MT(ASCP), Principal Investigator — Ingalls Memorial Hospital
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States